CLINICAL TRIAL: NCT00718796
Title: Naturopathic Treatment for the Prevention of Cardiovascular Disease: a Pragmatic Randomized Controlled Trial
Brief Title: Naturopathic Treatment for the Prevention of Cardiovascular Disease
Acronym: Cardio pilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Canada Post Corporation (Unknown); Canadian Union of Postal Workers (Other)
Responsible Party: Dugald Seely, Canadian College of Naturopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CP/CUPW4
Record Dates: First submitted 2008-04-25; First posted 2008-07-21 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular disease; naturopathic medicine; natural health products; lifestyle intervention; dietary advice; coronary heart disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease | interventions — Phytosterols; coenzyme Q10; Exercise; Diet; Complementary Therapies; Fish Oils; Atorvastatin; Anticholesteremic Agents; Fluvastatin; Lovastatin; Pravastatin; Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Individualized naturopathic treatment consisting of dietary and lifestyle advice and individualized supplementation
  Interventions: Other: Naturopathic medicine. May include: fish oil, plant sterols, soluble fiber, cinnamon, coQ10 and exercise
- 2 (Active Comparator): Current care control provided by participants' medical doctor
  Interventions: Other: Conventional medical treatment (Atorvastatin,Fluvastatin,Lovastatin,Pravastatin,Rosuvastatin,Simvastatin)

INTERVENTIONS:
Other: Naturopathic medicine. May include: fish oil, plant sterols, soluble fiber, cinnamon, coQ10 and exercise — Individualized according to needs of each participant and willingness to comply. Intervention to include lifestyle modification, dietary changes and supplementation using natural health products as recommended by naturopathic practitioner.
  Other Names: Naturopthic Medicine; Diet; Natural Health Products; Alternative Medicine; Fish oil; Plant sterols; Soluble fiber; CoQ10; Cinnamon; Exercise
  Arms: 1
Other: Conventional medical treatment (Atorvastatin,Fluvastatin,Lovastatin,Pravastatin,Rosuvastatin,Simvastatin) — Will vary according to individual - not standardized and likely to include statins.
  Other Names: Cholesterol lowering drugs; Atorvastatin; Fluvastatin; Lovastatin; Pravastatin; Rosuvastatin; Simvastatin
  Arms: 2

SUMMARY:
This study is designed to test the ability of a comprehensive naturopathic approach to reduce important risk factors for the development of cardiovascular disease. Treatment will take place over the course of one year and the comparator/control group will be followed by their medical doctors and be given conventional care.

DETAILED DESCRIPTION:
Interventions will consist of an individualized treatment approach guided by an expert panel of clinicians who treat patients with cardiovascular disease. These interventions will consist of a combination of dietary, lifestyle and specific recommendations for supplementation. As this is a pragmatic study, blinding will not be attempted nor is appropriate.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* CUPW worker
* prescreening indicates higher than normal TC/HDL ratio

Exclusion Criteria:

* Experienced an MI or stroke within past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome | 1 year
General Cardiovascular Risk Profile: Framingham Heart Study | 1 year

SECONDARY OUTCOMES:
Adverse events | 1 year
HbA1C | 1 year
Compliance with naturopathic interventions | 1 year
Quality of Life (Short-form 36) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dugald Seely, ND, Principal Investigator — Canadian College of Naturopathic Medicine
Locations (1):
- Canadian College of Naturopathic Medicine, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Herman PM, Szczurko O, Cooley K, Seely D. A naturopathic approach to the prevention of cardiovascular disease: cost-effectiveness analysis of a pragmatic multi-worksite randomized clinical trial. J Occup Environ Med. 2014 Feb;56(2):171-6. doi: 10.1097/JOM.0000000000000066. PMID 24451612
- [Derived] Seely D, Szczurko O, Cooley K, Fritz H, Aberdour S, Herrington C, Herman P, Rouchotas P, Lescheid D, Bradley R, Gignac T, Bernhardt B, Zhou Q, Guyatt G. Naturopathic medicine for the prevention of cardiovascular disease: a randomized clinical trial. CMAJ. 2013 Jun 11;185(9):E409-16. doi: 10.1503/cmaj.120567. Epub 2013 Apr 29. PMID 23630244
- See also: Central facility website — http://www.ccnm.edu